CLINICAL TRIAL: NCT00253058
Title: Evaluation of the Efficacy and Safety of Cetirizine Dry Syrup in Children -Suffering From Perennial Allergic Rhinitis-
Brief Title: Study Of Perennial Allergic Rhinitis In Pediatrics
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 104912
Record Dates: First submitted 2005-11-11; First posted 2005-11-15 (Estimated); Last update posted 2013-05-06 (Estimated); Status verified 2013-05

CONDITIONS: Rhinitis, Allergic, Perennial
Keywords: Allergic; pediatric; Rhinitis; Perennial
MeSH Terms: conditions — Rhinitis, Allergic, Perennial; Rhinitis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Cetirizine Dry Syrup

SUMMARY:
To verify of cetirizine dry syrup to ketotifen dry syrup in the change of total nasal symptom score (TNSS) over the total treatment period from the score of the baseline assessment period

ELIGIBILITY:
Inclusion Criteria:

* Children with perennial allergic rhinitis.
* Giving informed consent.
* Children with a positive response to specific IgE antibody test.
* Children assessed as positive in the nasal eosinophil count.
* Children whose severity score of nasal symptom is 4 or higher.

Exclusion criteria:

* have spastic disease such as epilepsy
* have a history of drug hypersensitivity
* are pregnant, lactating or possibly pregnant female Children
* are sensitive to pollen as a duplicate allergen and whose treatment periods are thought in the pollen dispersion periods
* have vasomotor rhinitis and eosinophilic rhinitis
* have asthma that requires the treatment with corticosteroid
* have inappropriate complication of nasal disorder that may influence on the evaluation of the study drugs
* have complicated with atopic dermatitis or urticaria that requires the treatment with antihistamine preparation
* have started specific desensitization treatment or nonspecific modulation treatment but who have not reached the maintenance level of treatment
* have received surgical treatment for reduction and modulation of nasal mucosa
* redintegration therapy of nasal cavity to improve the degree of nasal airway
* surgical operation to improve rhinorrhea.

Ages: 3 Years to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 286
Dates: Start 2005-07

PRIMARY OUTCOMES:
change in the total nasal symptom score (TNSS)

SECONDARY OUTCOMES:
- Individual daily nasal symptom score - Investigator global improvement/patient global improvement - Nasal findings - Cetirizine serum concentrations - Adverse events

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site